CLINICAL TRIAL: NCT04410731
Title: CellKine: Phase I Study Evaluating the Safety and Feasibility of Allogeneic, Culture-Expanded Bone Marrow-Derived Mesenchymal Stem Cells in Subjects with Painful Lumbar Facet Joint Arthropathy
Brief Title: Allogeneic BM-MSCs in Patients with Lumbar Facet Arthropathy
Acronym: Cellkine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wenchun Qu, Associate Professor of Anesthesiology and Physical Medicine and Rehabilitation, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-000330
Record Dates: First submitted 2020-05-14; First posted 2020-06-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Facet-Mediated Low Back Pain
Keywords: lumbar pain; facet joint; arthropathy
MeSH Terms: conditions — Low Back Pain; Joint Diseases

STUDY DESIGN:
Intervention Model Description: Staggered enrollment for subjects 1 to 3, followed by conditioned open enrollment for subjects 4 to 10.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BM-MSC injections for low back pain (Experimental): Single bilateral intra-articular injections of allogeneic BM-MSCs for lumbar facet joint arthropathy
  Interventions: Drug: Single bilateral intra-articular injection of allogeneic BM-MSCs for lumbar facet joint arthropathy

INTERVENTIONS:
Drug: Single bilateral intra-articular injection of allogeneic BM-MSCs for lumbar facet joint arthropathy — Single bilateral intra-articular injection of manufactured cell cultured expanded allogeneic BM-MSCs for painful lumbar facet joint arthropathy

SUMMARY:
Researchers are conducting this study to learn more about the side effects of bone marrow-derived stem cells when injected into the facet joints for the treatment of painful lumbar facet joint arthropathies.

DETAILED DESCRIPTION:
Phase I prospective study to determine the safety and feasibility of allogeneic, culture-expanded BM-MSCs in subjects with painful facet-mediated low back pain. Target accrual is 10 subjects with diagnosis of painful lumbar facet joint arthropathy. Eligible subjects will receive a single set of intra-articular bilateral injections of allogeneic, culture-expanded BM-MSCs human, allogeneic, culture expanded, bone-marrow-derived mesenchymal stem cells. Subjects will be evaluated at baseline, treatment day 0, post-operative day 1, post-operative days 3-5, week 2, and months 3, 6, 12, 18 and 24 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects ages 40-70 years who fulfill the following criteria:

1. Persons of childbearing potential must be non-nursing and have a negative serum pregnancy test to be included in the trial and will agree to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 24 months following completion of the drug treatment cycle.
2. Clinical diagnosis of symptomatic facet joint arthropathy involving the L3-S1 facets.
3. Radiographic evidence of facet arthropathy involving the L3-S1 facets.
4. Chronic low back pain with or without referred pain to the buttock, groin, or proximal thigh.
5. Confirmation of facet joint related pain by medial branch block with positive results.
6. Full understanding of the requirements of the study and willingness to comply with the treatment plan, including laboratory tests, diagnostic imaging, and follow-up visits and assessments.
7. Can provide written informed consent.

Exclusion Criteria:

1. Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI > 40)
2. Subjects who are pregnant or nursing or subjects planning to become pregnant in the first 24 months post-treatment.
3. Subjects with current or prior history of spinal infection at the symptomatic level.
4. Subjects with a diagnosis of severe osteoporosis with pathological fracture.
5. Radiofrequency ablation at the index level prior to injection in the past 3 months with positive results.
6. Any lumbar facet intra-articular injection including steroids at the index facet level prior to treatment injection in the past 3 months
7. Subjects that have undergone a procedure affecting the structure/biomechanics of the index facet joint or a spinal fusion adjacent to the symptomatic level.
8. Have undergone any procedure using biological treatment for any condition such as bone marrow aspirate concentrate, PRP, bone marrow-derived MSCs, adipose-derived MSCs, SVF, micro fragmented fat, embryonic membrane product etc.
9. Clinically relevant instability on flexion-extension as determined by the primary investigator by overlaying films.
10. Have an acute fracture of the spine at the time of enrollment in the study or clinically compromised vertebral bodies at the affected level due to current or past trauma.
11. Presence of any of the following spinal deformities: spondylolysis at the corresponding facet level, spondylolisthesis > grade II at the index facet.
12. Epidural steroid injections within 4 weeks prior to treatment injection.
13. Active malignancy or tumor as a source of symptoms or history of malignancy within the 5 years prior to enrollment in the study, except history of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or squamous cell carcinoma of the cervix if fully excised and with clear margins.
14. An elevated average baseline morphine equivalent dose, as determined by the investigator during screening consultation.
15. Taking systemic immunosuppressant medications or having a chronic, immunosuppressive state.
16. Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment.
17. Clinically significant abnormal hematology.
18. Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis.
19. Unexplained fever, defined as greater than 100.4 degrees Fahrenheit or 38.0 degrees Celsius, or mental confusion at baseline.
20. Clinically significant cardiovascular, neurological, renal, hepatic or endocrine disease.
21. Participation in a study of an experimental drug or medical device for treatment of facet joint arthropathy within one year.
22. Any contraindication to MRI according to MRI guidelines or unwillingness to undergo fluoroscopic procedures.
23. History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or medical marijuana
24. Any illness or condition which, in the investigators' judgment will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.
25. Being involved in active litigation related to subject's low back pain.
26. Have a mental illness that could prevent completion of the study or protocol questionnaires.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of nature, incidence, and severity of adverse events (AEs) | 24 months
  Clinical examination face-to-face during follow-up visits
Self-reported assessment of nature, incidence, and severity of AEs | 24 months
  Spontaneous subject reports
Study personnel assessment of nature, incidence, and severity of AEs | 24 months
  Subject interview by study personnel

SECONDARY OUTCOMES:
Global Health Scale (GHS) | 24 months
  Self-reported questionnaire to assess an individual's physical, mental, and social health. Standardized response scores ranges vary from1 to 5 (e.g., 1= None to 5=Very severe) or reversed (5=None to 1=Very severe) to ensure that higher scores for responses always indicate better health.
Visual Analog Scale (VAS) - back and leg pain | 24 months
  Subjective self-reported scale (1-10) to measure acute and chronic pain. (0= no pain; 10= worst pain possible).
Oswestry Disability Index (ODI) | 24 months
  Self-reported index to quantify disability for low back pain. Scores vary from 0 (no back pain) to 5 (worst back pain) in 10 sections (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). ODI Index is calculate.
Patient Health Questionnaire-4 (PHQ-4) | 24 months
  Self-reported brief questionnaire to screen for anxiety and depression. Four questions scoring 0 (not at all) to 3 (nearly every day).
Narcotic Use Questionnaire | 24 months
  Self-reported questionnaire to assess narcotic intake. Four questions to record narcotic drug usage (yes or no), frequency and length.
Work Status Questionnaire | 24 months
  Self-reported short questionnaire to assess work status at present. Simple 3 questions to record ability to work and to attend to work.
PROMIS-CAT | 24 months
  Patient-Reported Outcomes Measurement Information System to evaluate and monitor physical, mental, and social health. Standardized response scores ranges vary from1 to 5 (e.g., 1= None to 5=Very severe) or reversed (5=None to 1=Very severe) to ensure that higher scores for responses always indicate better health.
Changes from Baseline evaluated by MRI | 24 months
  Imaging evaluation by 2 independent radiographic interpretations to determine presence of effusions, bone marrow lesions/peri-articular edema, osteophytes, or any degree of facet synovitis
Change in number of red blood cells following treatment | 24 months
  Blood will be drawn in order to monitor for markers of systemic inflammation. The normal range of red blood cells varies slightly between laboratories but is generally between 4.2 - 5.9 million cells/cmm. This can also be referred to as the erythrocyte count and can be expressed in international units as 4.2 - 5.9 x 10^12 cells per liter.
Change in white blood cells with differential following treatment | 24 months
  Serological test - Automated white cell differential. A machine generated percentage of the different types of white blood cells, usually split into granulocytes, lymphocytes, monocytes, eosinophils, and basophils.
Change in number of platelets following treatment | 24 months
  Serological test: Platelets are not complete cells, but actually fragments of cytoplasm from a cell found in the bone marrow called a megakaryocyte. Platelets play a vital role in blood clotting. Normal range varies slightly between laboratories but is in the range of 150,000 - 400,000/ cmm (150 - 400 x 10^9/liter).
Change in Serum C-Reactive Protein (CRP) | 24 months
  Serological test: C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation throughout the body. It is one of a group of proteins called acute phase reactants that go up in response to inflammation. C-reactive protein is measured in milligrams of CRP per liter of blood (mg/L). Normal CRP levels are below 3.0 mg/dL.
Change in Erythrocyte Sedimentation Rate (ESR) | 24 months
  Serological test. The erythrocyte sedimentation rate (ESR) is the rate at which red blood cells sediment in a period of one hour. It is a common hematology test, and is a non-specific measure of inflammation. The normal range is 0-22 mm/hr for men and 0-29 mm/hr for women.
Change in Blood Urea Nitrogen (BUN) | 24 months
  Serological test - basic metabolic panel. A blood urea nitrogen (BUN) test measures the amount of nitrogen in the blood that comes from the waste product urea. Urea is made when protein is broken down in the body. Urea is made in the liver and passed out of the body in the urine. A BUN test is done to see how well the kidneys are working. Results of the blood urea nitrogen test are measured in milligrams per deciliter (mg/dL).
Change in Creatinine | 24 months
  Serological test - basic metabolic panel. Creatinine is a waste product produced by muscles from the breakdown of a compound called creatine. Almost all creatinine is filtered from the blood by the kidneys and released into the urine, so blood levels are usually a good indicator of how well the kidneys are working. Results are reported in mg/dL.
Change in Sodium | 24 months
  Serological test - basic metabolic panel. A sodium blood test allows the doctor to see how much sodium is in the subject's blood. It helps maintain normal blood pressure, supports the work of your nerves and muscles, and regulates your body's fluid balance. A normal sodium level is between 135 and 145 milliequivalents per liter (mEq/L) of sodium.
Change in Potassium | 24 months
  Serological test - basic metabolic panel. The normal potassium level in the blood is 3.5-5.0 milliEquivalents per liter (mEq/L).
Change in Chloride | 24 months
  Serological test - basic metabolic panel. The normal blood reference range of chloride for adults in most labs is 96 to 106 milliequivalents (mEq) per liter.
Change in Aspartate Aminotransferase (AST) | 24 months
  Serological test - basic metabolic panel. Inflamed or injured liver cells leak higher than normal amounts of certain chemicals, including liver enzymes, into the bloodstream, which can result in elevated liver enzymes on blood tests. The reference range for aspartate aminotransferase (AST) is as follows: Males: 6-34 IU/L, Females: 8-40 IU/L.
Change in Glucose | 24 months
  Serological test - basic metabolic panel. For a subject without diabetes, a fasting blood sugar on awakening should be under 100 mg/dl.
Change in Carbon Dioxide | 24 months
  Serological test - basic metabolic panel. The normal range for carbon dioxide is 23 to 29 mEq/L (milliequivalent units per liter of blood).

CONTACTS AND LOCATIONS:
Overall Officials: Wenchun Qu, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qu W, Yan D, Durand NC, Wang Z, Lehman VL, Osborne MD, Stone JA, Miller DA, Gupta S, Engelberg-Cook E, Wiest EF, Witter DM, Siebenaler KA, Quinones-Hinojosa A, Zubair AC. Intra-articular delivery of allogeneic bone marrow derived mesenchymal stromal cells (BM-MSCs) for painful lumbar facet arthropathy: a phase I clinical trial. Stem Cell Res Ther. 2025 Oct 30;16(1):596. doi: 10.1186/s13287-025-04674-y. PMID 41163019